CLINICAL TRIAL: NCT04067271
Title: LUEbeck Registry of Intensive Care Patients - Characterization of the Patients Intestinal MICROBIOME
Acronym: LUERIC-M
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Dr. med. Tobias Graf, Principal Investigator, University of Luebeck
Other Study IDs: 19-019
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: ICU Patients
MeSH Terms: interventions — Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analyze changes in intestinal microbiome — Descriptive Analysis

SUMMARY:
The purpose of the current study is to analyze the effects of ICU-care on changes in microbiome and the influence of intestinal microbiome changes on short-term and long-term morbidity and mortality of ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* All patients receiving intensive medical care
* A written informed consent from the patient or two independent doctors or legal guardians.

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive treatment on ICU.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2024-03-18 (Estimated); Study Completion 2024-03-18 (Estimated)

PRIMARY OUTCOMES:
Modification of the microbiome | Day 0
  The modification of the microbiome using ribosomal 16 S DNA sequencing and clustering for Operational Taxonomic Units (OTU) and calculated Shannon Index

SECONDARY OUTCOMES:
ICU intensive care unit stay | Day 0
  Duration
Hospital stay | Month 12
  Duration
Hospital stay | Month 6
  Duration
Survival | Month 6
  To discharge
Survival | Month 12
  To discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Clinic II-UKSH Campus Lübeck, Lübeck, Schleswig-Holstein, Germany